CLINICAL TRIAL: NCT06920511
Title: Integrated biO-cooPErative Robotic plAtform for Virtual Cognitive-motor Training in Parkinson's Disease
Brief Title: Cognitive Rehabilitation With Virtual Reality in Parkinson Disease
Acronym: OPERA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Università Campus Bio-Medico di Roma (UCBM) (Unknown); Khymeia Group S.r.l. (Unknown)
Responsible Party: Principal Investigator, Anna Estraneo, MD- Responsabile della Sperimentazione, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Opera; PNRR - AGE-IT SPOKE 1 e SPOKE (Other Grant/Funding Number: Ministero dell'Università e della Ricerca (MUR))
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Desease; Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The OPERA study is designed as a single-group interventional study. All participants are enrolled into one group and receive the same intervention, a cognitive rehabilitation program using the PRoBio platform. There are no comparison groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Training with PRoBio in Parkinson's Disease (Experimental): Patients with Parkinson's Disease and Mild Cognitive Impairment will undergo a cognitive rehabilitation program using the PRoBio robotic platform. The intervention consists of 3 sessions per week (45 minutes each) for 4 weeks. The PRoBio system includes virtual reality exercises and real-time feedback based on motor and emotional responses.
  Interventions: Device: Cognitve rehabilitation with virtual reality and robotic arm

INTERVENTIONS:
Device: Cognitve rehabilitation with virtual reality and robotic arm — The intervention consists of a cognitive rehabilitation program using the PRoBio platform, a bio-cooperative robotic system integrating virtual reality and real-time multisensory feedback. The PRoBio platform includes a robotic arm (TIAGo), a virtual reality interface (VRRS), and sensors to monitor biomechanical, cognitive, and emotional parameters during training.
  Other Names: TIAGo; COMPACT VRRS; Robotic Bio-Cooperative Training; Virtual Reality Rehabilitation with PRoBio; PRoBio platform

SUMMARY:
The OPERA Clinical Study is an interventional, single-arm, open-label pilot clinical study that aims to evaluate the usability of an innovative bio-cooperative robotic platform (PRoBio) for cognitive rehabilitation in patients with Parkinson's Disease (PD) and Mild Cognitive Impairment (MCI). The study focuses on assessing the effectiveness and acceptability of the system in a pilot study involving patients undergoing a structured cognitive rehabilitation program.

PRoBio is an advanced rehabilitation platform that integrates the TIAGo robotic system, developed by PAL Robotics, with the VRRS COMPACT virtual reality rehabilitation system, designed by Khymeia. TIAGo is provided by a robotic arm and RGB-D camera that allow the collection of biomechanical and psychophysiological data, which are then used to personalize the treatment through the cognitive tasks provided by the VRRS COMPACT. The pilot study involves patients with PD-MCI, who will undergo a four-week rehabilitation program with ProBio, consisting of three weekly sessions of virtual cognitive training. The primary objective is to assess the usability and compliance of the system by evaluating user experience, ease of interaction, and engagement levels among both patients and rehabilitation professionals, as well as evaluating its ability to monitor biomechanical and psychophysiological parameters during treatment. This assessment will be conducted using a multimodal sensor system, which includes an RGB-D camera integrated into the UCBM TIAGo robot and wearable sensors designed to measure heart rate, respiratory rate, and galvanic skin response. The data collected through these sensors will be analyzed offline to personalize cognitive rehabilitation treatments in subsequent sessions. Additionally, the study aims to evaluate the accuracy and response times of patients while performing cognitive exercises, as recorded by the VRRS system. Furthermore, the study will explore the potential effects of PRoBio treatment on the cognitive functions of patients with Parkinson's Disease and Mild Cognitive Impairment (PD-MCI) as a possible future rehabilitation to include in the clinical practice.

DETAILED DESCRIPTION:
The pilot study will be conducted at two clinical centers, the Fondazione Don Carlo Gnocchi ONLUS sites in Sant'Angelo dei Lombardi (AV) and Florence (FI).

The first step involves obtaining informed consent from all participants. Following this, a baseline assessment (T0) will be carried out, including the collection of demographic and anamnesis data, as well as cognitive and psychological evaluations. These assessments will help confirm eligibility criteria and serve as a pre-treatment evaluation for enrolled patients. The assessment tools include the MDS-Unified Parkinson's Disease Rating Scale, the Parkinson's Disease Cognitive Rating Scale, the Stroop Color Word Test, the Trail Making Test (A and B), the Parkinson's Disease Questionnaire (PDQ-39), the 15-item Geriatric Depression Scale, and the Geriatric Anxiety Inventory.

Once baseline evaluations are completed, patients will begin a structured cognitive rehabilitation program using the ProBio platform, which integrates the UCBM TIAGo service robot with the VRRS COMPACT telerehabilitation system developed by Khymeia. The rehabilitation program will consist of three weekly sessions, each lasting 45 minutes, for a total duration of four weeks. The cognitive tasks and activities will be tailored to the individual patient's abilities to provide a personalized treatment plan aimed at improving specific cognitive functions. During the rehabilitation sessions, UCBM TIAGo will continuously monitor the patient's physical and emotional state, collecting data through advanced sensors and its integrated RGB-D camera. These data will be analyzed offline to adjust the complexity and intensity of exercises for subsequent sessions based on individual responses.

Throughout the treatment, several parameters will be recorded. The accuracy and response times in cognitive exercises will be documented in reports generated by the VRRS software. Biomechanical parameters, such as movement amplitude and speed, will be measured using the RGB-D camera, while psychophysiological parameters, including respiratory rate, heart rate, and skin conductance, will be monitored via wearable sensors. Based on these parameters, the VRRS system will provide real-time visual and vocal feedback to the patient regarding response accuracy and exercise execution. Additionally, at the end of each session, the bio-cooperative robot TIAGo will verbally interact with the patient to assess their experience, including perceived enjoyment, task comprehension, and ease of execution.

At the end of the four-week rehabilitation program, a final evaluation (T1) will be conducted using the same cognitive and psychological assessment tools applied at baseline. This will include the MDS-Unified Parkinson's Disease Rating Scale, the Parkinson's Disease Cognitive Rating Scale, the Stroop Color Word Test, the Trail Making Test, the Parkinson's Disease Questionnaire (PDQ-39), the 15-item Geriatric Depression Scale, and the Geriatric Anxiety Inventory. The study also aims to explore the potential of integrating robotic bio-cooperative platforms into routine clinical rehabilitation settings, providing insights into their feasibility and effectiveness for future large-scale applications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild Parkinson's Disease (Hoehn & Yahr stage II-III);
* Diagnosis of Mild Cognitive Impairment (MCI) according to Litvan et al. (2012) criteria for PD-MCI;
* Age ≥ 18 years;
* Signed informed consent

Exclusion Criteria:

* Diagnosis of Parkinson's Disease Dementia, atypical parkinsonisms, secondary parkinsonisms, or mixed forms;
* Severe depressive syndrome
* Absence of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (SUS) - Patient Reported Outcome | Week 4 (post-treatment, T1)
  Assessment of system usability using the 10-item SUS scale. Scores range from 0 to 100; higher scores indicate better usability.
eHealth Usability Benchmarking Instrument (HUBBI) | Week 4 (post-treatment, T1)
  Assessment of system usability using the HUBBI questionnaire. Items rated on a 7-point scale; higher scores indicate better usability.
User Experience Questionnaire - Short Version (UEQ-S) | Week 4 (post-treatment, T1)
  Evaluation of pragmatic and hedonic user experience with the UEQ-S. Each item rated from -3 to +3; higher scores indicate more positive experience.
Technology Acceptance Model (TAM) and UTAUT Scores | Week 4 (post-treatment, T1)
  Evaluation of perceived usefulness and ease of use via TAM and UTAUT scales. Items rated on 5-point Likert scales.
NASA Task Load Index (NASA-TLX) | Week 4 (post-treatment, T1)
  Evaluation of cognitive workload using the NASA-TLX scale. Scores range from 0 to 100; higher scores indicate higher workload.

SECONDARY OUTCOMES:
Session Attendance and Treatment Adherence | Weeks 1-4
  Evaluation of the acceptance of the PRoBio platform by patients and clinicians, based on session attendance, treatment adherence, and system usability for operators. Additionally, the ability of PRoBio to collect biomechanical and psychophysiological data during treatment will be assessed. These include response accuracy and reaction times (collected by VRRS), movement amplitude and velocity (via RGB-D camera), and physiological indicators (heart rate, respiratory rate, and skin conductance) recorded through wearable sensors. These data will be used offline to customize the rehabilitation sessions.
Response Accuracy in Cognitive Tasks (VRRS Software) | Weeks 1-4
  Accuracy rate in exercises performed during each session, as recorded by VRRS.
Reaction Times in Cognitive Tasks (VRRS Software) | Weeks 1-4
  Mean reaction times (ms) recorded during cognitive tasks using the PRoBio platform.
Movement Amplitude (RGB-D Camera Analysis) | Weeks 1-4
  Mean amplitude of upper limb movements captured via RGB-D camera.
Movement Velocity (RGB-D Camera Analysis) | Weeks 1-4
  Mean velocity of arm movements during tasks, as measured by RGB-D camera.
Heart Rate During Sessions (Wearable Sensors) | Weeks 1-4
  Average heart rate recorded during rehabilitation sessions.
Respiratory Rate During Sessions (Wearable Sensors) | Weeks 1-4
  Average respiratory rate recorded during sessions.
Skin Conductance Level (SCL) During Sessions | Weeks 1-4
  Average SCL value measured by wearable sensors as indicator of emotional arousal.

OTHER OUTCOMES:
Cognitive Function - Parkinson's Disease Cognitive Rating Scale (PD-CRS) | Baseline (T0) and Week 4 (T1)
  PD-CRS scores will be collected to evaluate changes in cognitive performance. Scores range from 0 to 134; higher scores indicate better cognition.
Executive Function - Stroop Color Word Test (SCWT) | Baseline (T0) and Week 4 (T1)
  Performance on SCWT will be measured by response times and error rate.
Cognitive Flexibility - Trail Making Test (TMT A & B) | Baseline (T0) and Week 4 (T1)
  Completion time (in seconds) for TMT-A and TMT-B will be recorded.
Quality of Life - Parkinson's Disease Questionnaire (PDQ-39) | Baseline (T0) and Week 4 (T1)
  Quality of life will be measured through the PDQ-39. Scores range from 0 to 100; lower scores indicate better quality of life.
Mood - Geriatric Depression Scale (GDS-15) | Baseline (T0) and Week 4 (T1)
  Scores range from 0 to 15; higher scores indicate more depressive symptoms.
Anxiety - Geriatric Anxiety Inventory (GAI) | Baseline (T0) and Week 4 (T1)
  Scores range from 0 to 20; higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Estraneo, MD, Principal Investigator — Fondazione Don Gnocchi
Locations (1):
- Fondazione Don Gnocchi, Sant'Angelo dei Lombardi, Avellino, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared include demographic variables (age, gender, disease stage), usability and acceptability questionnaire scores, cognitive task performance (accuracy and reaction times), biomechanical parameters (e.g., movement amplitude and velocity), and psychophysiological data (e.g., heart rate, respiratory rate, skin conductance) collected during the intervention.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Access will be granted to qualified researchers affiliated with academic or clinical institutions, for the purpose of secondary analyses, meta-analyses, or method development. Requests must be submitted in writing to the principal investigator and will be evaluated by the study team. Data will be shared via secure file transfer methods upon approval.